CLINICAL TRIAL: NCT01965145
Title: A Randomized, Double-masked, Placebo-controlled Study of the Efficacy of Gevokizumab in the Treatment of Patients With Behçet's Disease Uveitis
Brief Title: Efficacy of Gevokizumab in the Treatment of Patients With Behçet's Disease Uveitis (EYEGUARD™-B)
Acronym: EYEGUARD™-B
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CL3-78989-002; 2012-001125-27 (EudraCT Number); U1111-1135-1411 (Other: WHO)
Record Dates: First submitted 2013-09-17; First posted 2013-10-18 (Estimated); Last update posted 2020-01-03 (Actual); Status verified 2020-01

CONDITIONS: Behcet's Uveitis
MeSH Terms: interventions — gevokizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gevokizumab (Experimental): Solution for subcutaneous injection, Dose 1
  Interventions: Drug: Gevokizumab
- Placebo (Placebo Comparator): Solution for subcutaneous injection, placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gevokizumab — Sterile solution administered subcutaneously
  Arms: Gevokizumab
Drug: Placebo — Sterile solution administered subcutaneously
  Arms: Placebo

SUMMARY:
The objective of this study is to demonstrate the superiority of gevokizumab as compared to placebo on top of current standard of care in reducing the risk of Behçet's disease uveitis exacerbations

DETAILED DESCRIPTION:
A randomized, double-masked, placebo-controlled study of the efficacy of gevokizumab in the treatment of patients with Behçet's disease uveitis

ELIGIBILITY:
Inclusion Criteria:

* Behçet's disease diagnosis fulfilling the International Study Group Classification Criteria.
* History of Behçet's disease uveitis with ocular involvement of the posterior segment.
* Patients with a stable background treatment of oral corticosteroid and at least one immunosuppressive drug.
* Male or female, age ≥18 (or legal age of majority in the country) at selection
* For subjects with reproductive potential, a willingness to use highly effective contraceptive measures

Exclusion Criteria:

* Infectious uveitis, uveitis due to causes other than Behçet's disease.
* Monocular vision
* Presence of severe cataract or severe posterior capsular opacification.
* Contraindication to mydriasis or presence of posterior synechiae.
* Active TB disease.
* History of severe allergic or anaphylactic reactions to monoclonal antibodies
* History of malignancy within 5 years prior to Selection.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2012-11; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Time to first acute ocular exacerbation | up to 3 years
  number of days

CONTACTS AND LOCATIONS:
Overall Officials: Sung Chul LEE, Pr, Principal Investigator — Severance Hospital
Locations (2):
- Yonsei University Severance Hospital, Seoul, South Korea
- St Thomas' Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Researchers can ask for a study protocol, patient-level and/or study-level clinical trial data including clinical study reports (CSRs).
  They can ask all interventional clinical studies:
  * submitted for new medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * Where Servier or an affiliate are the Marketing Authorization Holders (MAH). The date of the first Marketing Authorization of the new medicine (or the new indication) in one of the EEA Member States will be considered within this scope.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: http://clinicaltrials.servier.com

REFERENCES:
- [Result] Tugal-Tutkun I, Pavesio C, De Cordoue A, Bernard-Poenaru O, Gul A. Use of Gevokizumab in Patients with Behcet's Disease Uveitis: An International, Randomized, Double-Masked, Placebo-Controlled Study and Open-Label Extension Study. Ocul Immunol Inflamm. 2018;26(7):1023-1033. doi: 10.1080/09273948.2017.1421233. Epub 2018 Jan 25. PMID 29370572